CLINICAL TRIAL: NCT05112627
Title: Immunophenotyping in Metastatic Renal Cell Carcinoma Patients Receiving Ablative Therapy
Brief Title: Immunophenotyping in Metastatic Kidney Cancer Patients Receiving Ablative Therapy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley (Brad) Stish, Principal Investigator, Mayo Clinic
Other Study IDs: ROR2051; NCI-2021-10794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-011522 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-10-22; First posted 2021-11-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection): Patients undergo blood sample collection at baseline prior to SBRT or PCA, then at 14 days, 3 and 6 months after SBRT or PCA.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This early phase I trial evaluates blood samples to see if patients undergoing standard of care treatment with either stereotactic body radiation therapy or percutaneous ablation (using radio waves to create heat to destroy the tumor), have an increase in serum immune markers in kidney cancer. Information gained from this study may help doctors make treatment decisions for patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare pre- and post-treatment immune markers and peripheral blood mononuclear cell (PBMC) characteristics in metastatic renal cell carcinoma (RCC) patients overall.

II. Compare pre- and post-treatment immune markers and PBMC characteristics between patients being treated with stereotactic body radiation therapy (SBRT) versus percutaneous cryoablation (PCA) and are also undergoing immunotherapy.

III. Compare pre- and post-treatment immune markers and PBMC characteristics in patients being treated with either SBRT or PCA and not undergoing immunotherapy.

IV. Assess the impact of post-treatment immune markers and PBMC characteristics on distant disease progression in metastatic RCC patients overall.

OUTLINE:

Patients undergo blood sample collection at baseline prior to SBRT or PCA, then at 14 days, 3 and 6 months after SBRT or PCA.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary RCC
* Histological or radiographic diagnosis of metastatic RCC
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Feasible vascular access as determined by study staff
* Undergoing standard of care SBRT or PCA to RCC metastatic lesion(s)
* Provide written informed consent
* Willing to consent to research blood draws
* Willing to return to enrolling institution for follow-up

Exclusion Criteria:

* Prior local treatment of the index metastatic lesion
* Pregnant or nursing women
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for study entry
* Patients receiving prophylactic steroids, defined as initiation of steroids within 1 week prior to local ablative therapy start, including the first day of local ablative therapy.

  * NOTE: Patients initiating steroids after the first day of local ablative therapy and within 14 days after local ablative therapy completion, will be allowed into the study and the use of steroids will be recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological or radiographic diagnosis of metastatic RCC
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change in immune markers and peripheral blood mononuclear cell (PBMC) characteristics | Baseline up to 6 months
  Immune markers and PBMC characteristics will be evaluated overall. For change from baseline, comparisons between groups will be done using Analysis of Covariance (ANCOVA), including the pre-treatment count as a covariate in the model along with group status. The change will be described between groups reporting the mean and inter-quartile range. Linear regression will be used, analysis of covariance for change, for multiple variable models that will include any relevant baseline disease and patient characteristics.

SECONDARY OUTCOMES:
Change in immune markers and PBMC characteristics in patients undergoing stereotactic body radiation therapy (SBRT) versus percutaneous cryoablation (PCA) and receiving concurrent immunotherapy | Baseline up to 6 months
  Each CD8+ T cell will be compared between the SBRT and PCA groups using a two-sample T test at each of the time points as well as for percent change from baseline. For change from baseline, comparisons between groups will be done using ANCOVA, including the pre-treatment count as a covariate in the model along with group status. The change will be described between groups reporting the mean and inter-quartile range. Linear regression will be used, analysis of covariance for change, for multiple variable models that will include any relevant baseline disease and patient characteristics.
Change in immune markers and PBMC characteristics in patients undergoing SBRT or PCA and not receiving concurrent immunotherapy | Baseline up to 6 months
  Each CD8+ T cell will be compared between the SBRT and PCA groups using a two-sample T test at each of the time points as well as for percent change from baseline. For change from baseline, comparisons between groups will be done using ANCOVA, including the pre-treatment count as a covariate in the model along with group status. The change will be described between groups reporting the mean and inter-quartile range. Linear regression will be used, analysis of covariance for change, for multiple variable models that will include any relevant baseline disease and patient characteristics.
Levels of post-treatment immune markers and PBMC characteristics | Up to 6 months
  Will be correlated with distant disease progression overall (45 patients). Descriptive statistics will be used to summarize levels of immune markers and PBMC characteristics in the event of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Stish, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials